CLINICAL TRIAL: NCT05362565
Title: Genetic Research of Monogenic Obesity in a Pediatric Cohort With Severe and Early Onset Obesity
Acronym: OBEGENE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/55
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Monogenic Obesity
Keywords: monogenic obesity; pediatric; early onset obesity; genetic disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with salivary sampling
  Interventions: Biological: Salivary Sampling

INTERVENTIONS:
Biological: Salivary Sampling — The DNA study will be carried out from saliva sample
  1 saliva sample per patient will be performed at the inclusion visit

SUMMARY:
Obesity is a frequent disease mainly caused by environmental/polygenic factors and more rarely caused by the alteration of a single gene ("monogenic obesity"). The diagnosis of these rare forms can lead to personalized management (new treatments, prognosis, adapted hygienic and dietary rules) and family screening. The use of a panel covering the known causes of monogenic obesity on a pediatric cohort of severe and early obesity will allow to evaluate the relevance of these analyses to adapt the management of this type of patients.

ELIGIBILITY:
Inclusion Criteria:

* Recruitment age: 2-17 years
* Body mass index, greater than the International Obesity Task Force (IOTF) 30 curve before the age of 5
* Care at the specialized pediatric obesity center (CSO) of the Bordeaux University Hospital
* Informed consent signed

Exclusion Criteria:

* no informed consent

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient with a Body mass index, greater than the International Obesity Task Force (IOTF) 30 curve before the age of 5.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Positivity rate of patients for whom a diagnosis of monogenic obesity will be obtained when all analyses have been performed. | Inclusion visit

SECONDARY OUTCOMES:
Number of Patients eligible for a drug targeting single-gene obesity | Inclusion visit
Number of patients for whom a genetic finding will have changed management and description of changes. | Inclusion visit

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No